CLINICAL TRIAL: NCT03680105
Title: A Phase 1, Double-blind, Placebo-controlled, Randomized, Two-Part, Ascending Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Rejuveinix (RJX) in Healthy Participants
Brief Title: A Safety and Tolerability Study of RJX Drug Product in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reven Pharmaceuticals, Inc. (Industry)
Collaborators: ICON plc (Industry); ERT: Clinical Trial Technology Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RPI003
Record Dates: First submitted 2018-08-29; First posted 2018-09-21 (Actual); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1; Cohort 1; RJX or Placebo (Experimental): Participants in Part 1; Cohort 1 will receive a single 0.024 mL/kg dose of RJX or matching placebo on Day 1.
  Interventions: Drug: RJX; Drug: Placebo
- Part 1; Cohort 2; RJX or Placebo (Experimental): Participants in Part 1; Cohort 2 will receive a single 0.076 mL/kg dose of RJX or matching placebo on Day 1.
  Interventions: Drug: RJX; Drug: Placebo
- Part 1; Cohort 3; RJX or Placebo (Experimental): Participants in Part 1; Cohort 3 will receive a single 0.240 mL/kg dose of RJX or matching placebo on Day 1.
  Interventions: Drug: RJX; Drug: Placebo
- Part 1; Cohort 4; RJX or Placebo (Experimental): Participants in Part 1; Cohort 4 will receive a single 0.5 mL/kg dose of RJX or matching placebo on Day 1.
  Interventions: Drug: RJX; Drug: Placebo
- Part 1; Cohort 5; RJX or Placebo (Experimental): Participants in Part 1; Cohort 5 will receive a single 0.759 mL/kg dose of RJX or matching placebo on Day 1.
  Interventions: Drug: RJX; Drug: Placebo
- Part 1; Cohort 6; RJX or Placebo (Experimental): Participants in Part 1; Cohort 6 will receive a single dose of RJX or matching placebo, to be determined following review of safety and PK data from Cohorts 1 to 5, on Day 1.
  Interventions: Drug: RJX; Drug: Placebo
- Part 2; Cohort 1; RJX or Placebo (Experimental): Participants in Part 2; Cohort 1 will receive a dose of RJX or matching placebo, determined based on the findings of Part 1, every day for 7 days.
  The Part 2; Cohort 1 dose will be 1 log down from the maximum tolerated dose determined in Part 1 or at a dose determined to be safe and well tolerated in Part 1 with an acceptable PK profile.
  Interventions: Drug: RJX; Drug: Placebo
- Part 2; Cohort 2; RJX or Placebo (Experimental): Participants in Part 2; Cohort 2 will receive an escalated dose of RJX or matching placebo, determined based on the findings of Part 1, every day for 7 days.
  Interventions: Drug: RJX; Drug: Placebo
- Part 2; Cohort 3; RJX or Placebo (Experimental): Participants in Part 2; Cohort 3 will receive an escalated dose of RJX or matching placebo, determined based on the findings of Part 1, every day for 7 days.
  Interventions: Drug: RJX; Drug: Placebo

INTERVENTIONS:
Drug: RJX — RJX is an IV infusion formulation. The appropriate RJX dose is calculated based on mL/kg. The administration dose is prepared by adding the appropriate RJX dose to 0.9% sterile saline such that a constant volume of 100 mL per IV infusion is obtained. Infusion time is 100 mL over 45 minutes (+/- 5 minutes).
Drug: Placebo — Matching placebo will be normal saline. To maintain the blind, a sleeve will cover the infusion bag and line such that the appearance will be identical to RJX administration.

SUMMARY:
Designed as a single center, two-part, double-blind, placebo-controlled, randomized study to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of RJX in healthy participants.

DETAILED DESCRIPTION:
Part 1 is designed as a Single Ascending Dose (SAD) escalation study with 6 cohorts. Participants will undertake a screening visit between Day -21 and Day -1 to determine eligibility in the study. Those participants that meet the eligibility criteria will be admitted to the study site on the day prior to dosing (Day -1). Participants will receive a single dose of investigational product via IV infusion on Day 1. The first cohort will include the initial dosing of a sentinel group. The remaining participants in Cohort 1 will be dosed if, in the opinion of the investigator or delegate, there are no significant safety concerns identified in the sentinel participants within the first 24 hours after administration of the dose. Participants will be confined to the study site from Day -1 to Day 2 (24 hours post dose) and then required to return to the study site on Day 5 for a final follow up visit. Safety and PK assessments will be performed at selected time points throughout the study.

Part 2 is designed as a Multiple Ascending Dose (MAD) escalation study with 3 cohorts. The MAD arm of the study will commence in parallel with Cohort 6 of Part 1 following completion and review of safety and PK findings for Cohorts 1, 2, 3, 4, and 5 in Part 1. Participants will undertake a screening visit between Day -21 and Day -1 to determine eligibility in the study. Those participants that meet the eligibility criteria will be admitted to the study site on the day prior to dosing (Day -1). Participants will be randomly assigned to receive 1 of 3 proposed doses of investigational product via IV infusion every day for 7 days.Participants will be confined to the study site from Day -1 to Day 8 (24 hours post the final dose on Day 7) and then return to the study site on Day 12 for a final follow up visit. Safety and PK assessments will be performed at selected time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged 18 to 50 years inclusive (Cohort 1 to Cohort 5) or 51 to 70 years inclusive (Cohort 6 only),at the time of screening;
2. Have a body mass index of 18 kg/m2 to 35 kg/m2, inclusive, at screening. In addition, weight cannot exceed 132 kg;
3. Have negative screening assessment for viral hepatitis (hepatitis B or hepatitis C) and human immunodeficiency virus;
4. Have negative routine urine drug screen and negative alcohol breath test at screening and Day -1;
5. A female participant is eligible to participate if she is not pregnant,not breastfeeding, and at least 1 of the following conditions applies:

   1. Not of childbearing potential, defined as surgically sterile (documented hysterectomy, bilateral salpingectomy, tubal ligation or bilateral oophorectomy) or postmenopausal (no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient);
   2. Of childbearing potential and agrees to use 2 highly effective methods of contraception consistently during the treatment period and for at least 60 days after the last dose of investigational product;
6. A male participant with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception during the treatment period and for at least 60 days after the last dose of investigational product and refrains from donating sperm during this period;
7. Clinical laboratory test results within normal reference range for the population or investigator site, or any results that are judged to be not clinically significant by the investigator;
8. Venous access sufficient to allow for blood sampling per the protocol;
9. Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures;
10. Given written informed consent prior to any study procedures being performed

Exclusion Criteria:

1. Have a history of clinically relevant cardiovascular disease, cancer, respiratory, hepatic, renal, gastrointestinal, endocrine (diabetes), hematological, or neurological disorders. Cohort 6 only - elderly participants with well controlled hypercholesterolemia on a stable dose of statin therapy or well controlled hypertension on a stable dose of antihypertensive medication(s), excluding diuretics, are allowed in Cohort 6 per the clinical judgment of the investigator.
2. Have impaired renal function (defined as estimated glomerular filtration rate <90 cc/min/1.73m2 Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) creatinine equation at screening);
3. Have a hsCRP above 1.25 × upper limit of normal;
4. Have a clinically significant abnormality in the 12-lead electrocardiogram (ECG) or prolongation of corrected QT interval by Fredericia (QTcF) >440 ms in males and >450 ms in females;
5. Have a supine systolic blood pressure (BP) greater than 140 mm Hg or a diastolic BP greater than 90 mm Hg. Up to 2 additional measurements may be undertaken after an appropriate resting interval at screening to confirm eligibility;
6. Are currently enrolled in a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study;
7. Have received an investigational product within the last 3 months;
8. Have suspected allergies to RJX, related compounds, or any components of the formulation, or history of significant atopy;
9. Regularly use known drugs of abuse and/or show positive findings on drug screening or Day -1;
10. Are women who are pregnant, intend to become pregnant, or are lactating;
11. Participants will be excluded for using any of the following medication:

    * aspirin, multivitamins/vitamins or mineral preparations within 14 days prior to investigational product administration or 24 hours post the last infusion;
    * prescription, herbal or over the counter medications within 14 days of investigational product administration, with the exception of:

      * simple analgesics such as paracetamol, excluding aspirin
      * oral non-steroidal anti-inflammatory drugs
      * thyroid treatment, estrogen replacement therapy
      * hormonal contraception
      * Statins and anti-hypertensives are permitted for elderly participants in Cohort 6 (Part 1) - see inclusion criteria #1
12. Have donated blood of more than 500 mL within 4 weeks prior to study enrollment;
13. Have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females) or are unwilling to stop alcohol consumption for 24 hours prior to study site admission (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits). Participants must have a of negative alcohol breath test at Day -1 and no evidence of alcohol abuse in the previous 12 months, defined as > 21 weekly units for males up to age 65 and > 14 weekly units for males over 65 and females;
14. Have smoked cigarettes in the last 90 days (including occasional smokers who have smoked more than 5 cigarettes per month within the last 90 days);
15. In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study;
16. Are investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted;
17. Are Reven employees or employees of third-party organizations involved with the study who require exclusion of their employees.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis A Ruff, MD, Principal Investigator — ICON Early Phase Services
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

REFERENCES:
- [Derived] Uckun FM, Saeed M, Awili M, Ozercan IH, Qazi S, Lee C, Shibli A, Skolnick AW, Prusmack A, Varon J, Barrera CI, Orhan C, Volk M, Sahin K. Evaluation of the potential of Rejuveinix plus dexamethasone against sepsis. Future Microbiol. 2022 Oct;17:1217-1229. doi: 10.2217/fmb-2022-0044. Epub 2022 Sep 2. PMID 36052743
- [Derived] Uckun FM, Orhan C, Tuzcu M, Durmus AS, Ozercan IH, Volk M, Sahin K. RJX Improves Wound Healing in Diabetic Rats. Front Endocrinol (Lausanne). 2022 Jun 2;13:874291. doi: 10.3389/fendo.2022.874291. eCollection 2022. PMID 35721744
- [Derived] Uckun FM, Carlson J, Orhan C, Powell J, Pizzimenti NM, van Wyk H, Ozercan IH, Volk M, Sahin K. Rejuveinix Shows a Favorable Clinical Safety Profile in Human Subjects and Exhibits Potent Preclinical Protective Activity in the Lipopolysaccharide-Galactosamine Mouse Model of Acute Respiratory Distress Syndrome and Multi-Organ Failure. Front Pharmacol. 2020 Nov 10;11:594321. doi: 10.3389/fphar.2020.594321. eCollection 2020. PMID 33244300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants received either Rejuveinix (RJX) or saline placebo.
Groups:
- Part 1; Cohort 1; RJX or Placebo: Participants in Part 1; Cohort 1 received a single 0.024 mL/kg dose of RJX or matching placebo on Day 1.
- Part 1; Cohort 2; RJX or Placebo: Participants in Part 1; Cohort 2 received a single 0.076 mL/kg dose of RJX or matching placebo on Day 1.
- Part 1; Cohort 3; RJX or Placebo: Participants in Part 1; Cohort 3 received a single 0.240 mL/kg dose of RJX or matching placebo on Day 1.
- Part 1; Cohort 4; RJX or Placebo: Participants in Part 1; Cohort 4 received a single 0.500 mL/kg dose of RJX or matching placebo on Day 1.
- Part 1; Cohort 5; RJX or Placebo: Participants in Part 1; Cohort 5 received a single 0.759 mL/kg dose of RJX or matching placebo on Day 1.
- Part 1; Cohort 6; RJX or Placebo: Participants in Part 1; Cohort 6 received a single dose of 0.500 mL/kg RJX or matching placebo on Day 1.
  Cohort 6 subjects comprised a cohort of healthy volunteers aged 51-70 inclusive.
- Part 2; Cohort 1; RJX or Placebo: Participants in Part 2; Cohort 1 received a dose of 0.240 mL/kg RJX or matching placebo every day for 7 days.
- Part 2; Cohort 2; RJX or Placebo: Participants in Part 2; Cohort 2 received a dose of 0.500 mL/kg RJX or matching placebo every day for 7 days.
- Part 2; Cohort 3; RJX or Placebo: Participants in Part 2; Cohort 3 received a dose of 0.759 mL/kg RJX or matching placebo every day for 7 days.
Period: Overall Study
Arm/Group | Part 1; Cohort 1; RJX or Placebo | Part 1; Cohort 2; RJX or Placebo | Part 1; Cohort 3; RJX or Placebo | Part 1; Cohort 4; RJX or Placebo | Part 1; Cohort 5; RJX or Placebo | Part 1; Cohort 6; RJX or Placebo | Part 2; Cohort 1; RJX or Placebo | Part 2; Cohort 2; RJX or Placebo | Part 2; Cohort 3; RJX or Placebo
Started | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1; Cohort 1; RJX or Placebo | Part 1; Cohort 2; RJX or Placebo | Part 1; Cohort 3; RJX or Placebo | Part 1; Cohort 4; RJX or Placebo | Part 1; Cohort 5; RJX or Placebo | Part 1; Cohort 6; RJX or Placebo | Part 2; Cohort 1; RJX or Placebo | Part 2; Cohort 2; RJX or Placebo | Part 2; Cohort 3; RJX or Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8 | 76
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 5 | 3 | 7 | 0 | 4 | 5 | 39
  Male | 3 | 4 | 2 | 3 | 5 | 5 | 8 | 4 | 3 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 2 | 2 | 3 | 5 | 3 | 4 | 2 | 0 | 7 | 28
  White | 6 | 6 | 5 | 3 | 5 | 8 | 5 | 8 | 1 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8 | 76

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Adverse Events (TEAE) Reporting of RJX
Description: Number of participants with indicated AEs receiving RJX as assessed by CTCAE v4 03
Time Frame: Up to Day 5 for Part 1 and Up to Day 12 for Part 2
Measure: Count of Participants; unit: Participants
Groups:
- Part 1; Placebo: Participants in Part 1 received a single saline placebo on Day 1.
- Part 1; Cohort 1; RJX: Participants in Part 1; Cohort 1 received a single 0.024 mL/kg dose of RJX or matching placebo on Day 1.
- Part 1; Cohort 2; RJX: Participants in Part 1; Cohort 2 received a single 0.076 mL/kg dose of RJX on Day 1.
- Part 1; Cohort 3; RJX: Participants in Part 1; Cohort 3 received a single 0.240 mL/kg dose of RJX on Day 1.
- Part 1; Cohort 4; RJX: Participants in Part 1; Cohort 4 received a single 0.500 mL/kg dose of RJX on Day 1.
- Part 1; Cohort 5; RJX: Participants in Part 1; Cohort 5 received a single 0.759 mL/kg dose of RJX on Day 1.
- Part 1; Cohort 6; RJX: Participants in Part 1; Cohort 6 received a single dose of 0.500 mL/kg RJX Day 1.
  Cohort 6 subjects comprised a cohort of healthy volunteers aged 51-70 inclusive.
- Part 2; Placebo: Participants in Part 2 received a dose of saline placebo every day for 7 days.
- Part 2; Cohort 1; RJX: Participants in Part 2; Cohort 1 received a dose of 0.240 mL/kg RJX every day for 7 days.
- Part 2; Cohort 2; RJX: Participants in Part 2; Cohort 2 received a dose of 0.500 mL/kg RJX every day for 7 days.
- Part 2; Cohort 3; RJX: Participants in Part 2; Cohort 3 received a dose of 0.759 mL/kg RJX every day for 7 days.
Arm/Group | Part 1; Placebo | Part 1; Cohort 1; RJX | Part 1; Cohort 2; RJX | Part 1; Cohort 3; RJX | Part 1; Cohort 4; RJX | Part 1; Cohort 5; RJX | Part 1; Cohort 6; RJX | Part 2; Placebo | Part 2; Cohort 1; RJX | Part 2; Cohort 2; RJX | Part 2; Cohort 3; RJX
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 6
Participants
  Mild TEAE: With TEAE | 2 | 1 | 2 | 0 | 2 | 2 | 0 | 1 | 1 | 3 | 2
  Mild TEAE: Without TEAE | 11 | 5 | 4 | 6 | 4 | 4 | 9 | 5 | 5 | 3 | 4
  Moderate TEAE: With TEAE | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
  Moderate TEAE: Without TEAE | 13 | 6 | 6 | 6 | 5 | 5 | 9 | 5 | 6 | 6 | 5
  Severe TEAE: With TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe TEAE: Without TEAE | 13 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 6
  Related TEAE: With TEAE | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 0
  Related TEAE: Without TEAE | 13 | 5 | 5 | 6 | 4 | 4 | 9 | 5 | 6 | 4 | 6

2. Primary Outcome: Safety and Tolerability of RJX as Assessed by Electrocardiograms (ECGs).
Description: Number of participants with abnormal and clinically significant findings based on ECG.
Time Frame: Up to Day 2 for Part 1 and Up to Day 8 for Part 2
Population: Counts of 12-lead safety ECG interpretations across Intent to Treat (ITT) population showed no notable changes when compared to baseline for either study part.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1; Placebo | Part 1; Cohort 1; RJX | Part 1; Cohort 2; RJX | Part 1; Cohort 3; RJX | Part 1; Cohort 4; RJX | Part 1; Cohort 5; RJX | Part 1; Cohort 6; RJX | Part 2; Placebo | Part 2; Cohort 1; RJX | Part 2; Cohort 2; RJX | Part 2; Cohort 3; RJX
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Safety and Tolerability of RJX as Assessed by Neurological Examinations.
Description: Number of participants with clinically significant values and actual changes from baseline of continuous neurological assessments.
Time Frame: Up to Day 5 for Part 1 and Up to Day 12 for Part 2
Population: Analysis based on Intent to Treat (ITT) population across Part 1 and Part 2, all cohorts. Only 1 subject, one incidence, for the study; presented on Day 12, Principal Investigator considered clinically significant and a mild TEAE considered unlikely related to RJX.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1; Placebo | Part 1; Cohort 1; RJX | Part 1; Cohort 2; RJX | Part 1; Cohort 3; RJX | Part 1; Cohort 4; RJX | Part 1; Cohort 5; RJX | Part 1; Cohort 6; RJX | Part 2; Placebo | Part 2; Cohort 1; RJX | Part 2; Cohort 2; RJX | Part 2; Cohort 3; RJX
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Part 1 (SAD): 5 Days Part 2 (MAD) 12 Days
Groups:
- Part 1; Cohort 1; RJX: Participants in Part 1; Cohort 1 received a single 0.024 mL/kg dose of RJX on Day 1.
- Part 1; Cohort 6; RJX: Participants in Part 1; Cohort 6 receive a single dose of 0.500 mL/kg RJX on Day 1.
  Cohort 6 subjects comprised a cohort of healthy volunteers aged 50-70 inclusive.
- Part 2; Placebo: Participants in Part 2 received a saline placebo every day for 7 days.
- Part 2; Cohort 2; RJX or Placebo: Participants in Part 2; Cohort 2 received a dose of 0.500 mL/kg RJX every day for 7 days.
- Part 2; Cohort 3; RJX or Placebo: Participants in Part 2; Cohort 3 received a dose of 0.759 mL/kg RJX every day for 7 days.
Arm/Group | Part 1; Placebo | Part 1; Cohort 1; RJX | Part 1; Cohort 2; RJX | Part 1; Cohort 3; RJX | Part 1; Cohort 4; RJX | Part 1; Cohort 5; RJX | Part 1; Cohort 6; RJX | Part 2; Placebo | Part 2; Cohort 1; RJX | Part 2; Cohort 2; RJX or Placebo | Part 2; Cohort 3; RJX or Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/13 | 1/6 | 2/6 | 0/6 | 3/6 | 2/6 | 0/9 | 1/6 | 1/6 | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1; Placebo (N=13) | Part 1; Cohort 1; RJX (N=6) | Part 1; Cohort 2; RJX (N=6) | Part 1; Cohort 3; RJX (N=6) | Part 1; Cohort 4; RJX (N=6) | Part 1; Cohort 5; RJX (N=6) | Part 1; Cohort 6; RJX (N=9) | Part 2; Placebo (N=6) | Part 2; Cohort 1; RJX (N=6) | Part 2; Cohort 2; RJX or Placebo (N=6) | Part 2; Cohort 3; RJX or Placebo (N=6)
Infusion site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delayed Sleep Phase (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Ankle clonus
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Systolic Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive Protein Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT03680105/Prot_SAP_000.pdf